CLINICAL TRIAL: NCT05547620
Title: Modulating Dysfunctional Cerebellar Activity With Low-intensity Focused Ultrasound Stimulation for Primary Orthostatic Tremor
Brief Title: Modulating Cerebellar Activity With Low-intensity Focused Ultrasound Stimulation for Primary Orthostatic Tremor
Acronym: LIFUS-POT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Organization for Rare Disorders (Other)
Responsible Party: Principal Investigator, Robert Chen, Senior Scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-5740
Record Dates: First submitted 2022-03-03; First posted 2022-09-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Orthostatic Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low Intensity Focused ultrasound (Experimental): NeuroFUS device stimulation with 4 channel transducer Stimulation target = Cerebellum
  Interventions: Device: LIFUS Online Real; Device: LIFUS Online Sham; Device: LIFUS Offline

INTERVENTIONS:
Device: LIFUS Online Real — Stimulation using NeuroFUS device while standing
Device: LIFUS Online Sham — Stimulation using NeuroFUS device while standing
Device: LIFUS Offline — Stimulation using NeuroFUS device prior to standing

SUMMARY:
Primary orthostatic tremor (POT) is a rare movement disorder that is manifested through high frequency tremor of weight bearing limbs. This is often accompanied by a debilitating sensation of falling. POT has been linked to abnormal activity of the cerebellum, a structure deep within the brain. However, established non-invasive brain stimulation techniques can only modulate brain activity and plasticity in superficial brain areas with low spatial resolution. This limits their efficacy when targeting the cerebellum. In contrast, low intensity focused ultrasound (LIFUS) is a novel non-invasive brain stimulation technique that permits stimulation with high spatial focality and can reach greater depth compared other methods. Therefore, LIFUS is well suited to modulate cerebellar activity and has the potential to be a superior technique for the management of POT. This study will investigate the effectiveness of MRI-guided bilateral cerebellar LIFUS stimulation for the treatment of POT and evaluate the underlying changes in brain circuits caused by the stimulation. Comparisons between symptoms and connectivity of brain circuits pre- and post-stimulation will be conducted to assess the effects of cerebellar LIFUS. The effects of real stimulation will also be compared to sham stimulation. This study is the first to apply LIFUS for neuromodulation in POT and will be critical in developing therapeutic LIFUS protocols.

DETAILED DESCRIPTION:
In the current study the investigators aim to assess the effects of low intensity focused ultrasound (LIFUS) on the symptoms of primary orthostatic tremor (POT) and on brain connectivity. LIFUS is a promising non-invasive brain stimulation technique that is actively being studied for its ability to reversibly modulate brain activity. By focusing the propagation of acoustic wave through the skull, a higher degree of spatial specificity and deep targeting can be achieved over other non-invasive stimulation methods such as transcranial magnetic stimulation (TMS) and transcranial direct-current stimulation (tDCS). Specifically, investigators will use LIFUS to stimulate the cerebellum bilaterally for 80s per hemisphere using a theta burst protocol that investigators have shown to induce plasticity. Investigators hypothesize that modulating cerebellar activity will decrease symptoms of POT and normalize the dysfunctional cerebello-thalamo-cortico network. 15 POT patients will be recruited to participate in 3 sessions in-lab. The first visit will involve an anatomical magnetic resonance image (MRI) scan. This will allow us to accurately target cerebellar lobule VIII and establish the appropriate parameters of LIFUS to effectively pass through the skull. In visits 2 and 3 participants will be seated in a comfortable chair and an anatomical MRI image will be used to position the LIFUS transducer over cerebellar lobule VIII bilaterally on surface of their head. In visit 2, clinical assessments of POT will be conducted through electromyography (EMG) recordings and video analysis of posture and sway. Symptoms prior to and after LIFUS will be compared. Investigators will compare the effects of real stimulation to a sham stimulation. In visit 3, Investigators will assess brain network activity using transcranial magnetic stimulation (TMS) by employing an established paired-pulse paradigm. This method will allow us to establish the effects of LIFUS on the cerebello-thalamo-cortical network and determine how this related to changes observed in POT symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years of age
* Confirmed diagnosis of orthostatic tremor

Exclusion Criteria:

* History of stroke or seizure
* Comorbid dementia
* Scored below 22 on the Montreal Cognitive Assessment (MoCA)
* Has intracranial implant(s) or device(s)
* Has an implanted cardiac pacemaker or implantable cardioverter-defibrillator (ICD)
* Has a previous surgical intervention to treat the movement disorder such as lesioning or a deep brain stimulation (DBS) system in place.
* Presence of metal implanted in body that is contraindicated in TMS/MRI
* Pregnancy
* Major depression/psychiatric disorder that in the opinion of the Investigator will affect patient's understanding of study procedures and willingness to abide by all procedures during the course of the study
* Is on antipsychotics, marijuana, or other recreational drugs that affect the nervous system
* Major musculoskeletal or neuromuscular disease or disorder of the hands, wrists and limbs
* Major systemic illness or infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Tremor frequency | 2 Years
  The primary outcomes will consist of peak tremor frequency recorded from surface electromyography (EMG). The EMG electrodes will be placed on the skin, and electrical activity produced by muscle contractions will be recorded. From the recordings of EMGs, peak frequency will be extracted through statistical analyses.
Power spectral analysis | 2 Years
  Power spectrum recorded from surface electromyography (EMG). The EMG electrodes will be placed on the skin, and electrical activity produced by muscle contractions will be recorded. From the recordings of EMGs, power spectrum will be extracted through statistical analyses.
Orthostatic Tremor Severity and Disability Scale (OT-10) | 2 Years
  The Orthostatic Tremor Severity and Disability Scale (OT-10) is a self-administered 10-item scale that measures the severity and disability of orthostatic tremor. Each item is rated from 0-5, with higher scores representing worse outcome.

SECONDARY OUTCOMES:
Assessment of body posture | 2 Years
  Posture during standing will be video recorded and analyzed using Kinovea, an analysis software for evaluation of human movements that express measurements in figures, tables, and graphics. Specifically, posture analysis will be carried out by measuring the alignment of the head, shoulder, hips, knees, and ankles. Deviation scores for each alignment measure will be calculated and averaged to calculate an overall alignment deviation score for each participant.
Standing time | 2 Years
  Duration of standing

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, MBBS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No